CLINICAL TRIAL: NCT05073952
Title: Width of Keratinazed Mucosa in Immediately Loaded Posterior Implant Restorations Treated With Different Surgical Approaches: Randomized Clinical Study.
Brief Title: Keratized Mucosa in CG Implant Placement: CTG vs Flapless
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Milan (Other)
Responsible Party: Principal Investigator, Stefano Storelli, Reasearcher, University of Milan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: KM001
Record Dates: First submitted 2021-09-17; First posted 2021-10-12 (Actual); Last update posted 2021-12-03 (Actual); Status verified 2021-12

CONDITIONS: Variation of Keratinized Mucosa After Implant Surgery
Keywords: dental implant; Keratinized mucosa; Connective tissue graft; flapless implant placement; Computer guided implantology; Immediate loading

STUDY DESIGN:
Intervention Model Description: two groups will be compared with different treatment
Who Masked: Outcomes Assessor
Masking Description: surgical treatment will be conducted with surgeon-investigator and patient unblinded. the outcome assessor will be blinded as primary outcome measurements will be taken on a computer.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Connective tissue graft (Active Comparator): patient in this group will be treated with a flap and a connective tissue graft at the moment of implant placement.
  Interventions: Procedure: Connective tissue graft
- Flapess (Active Comparator): patient in this group will be treated with a flapless approach at the moment of implant placement.
  Interventions: Procedure: Flapless

INTERVENTIONS:
Procedure: Connective tissue graft — Implants will be placed with a flap and a connective tissue graft.
  Arms: Connective tissue graft
Procedure: Flapless — Implants will be placed with a flapless approach
  Arms: Flapess

SUMMARY:
The present study will evaluate the difference in terms of keratinazed mucosa (KM) in computer guided implant placement with immediate loading, comparing a flapless approach to flap surgery with connective tissue graft.

ELIGIBILITY:
Inclusion Criteria:

* Age 18+
* Patients with partial edentulism in the posterior region (4-7) upper or lower for at least 3 months
* Patient whose tomographic examination shows adequate bone volumes for computer guided placement of a standard diameter implant (> 3.5 mm) without the need for bone regeneration procedures
* Patients who have accepted informed consent and participation in the study
* Patients who do not have exclusion criteria

Eclusion Criteria

* Patients who refuse to co-operate
* Systemic conditions of exclusion:

  * Medical conditions requiring prolonged use of steroids
  * Severe hemophilia
  * In therapy with intravenous bisphosphonates
  * History of white blood cell dysfunction or deficiency
  * History of head and neck radiotherapy or chemotherapy
  * History of kidney failure
  * Pregnant or breastfeeding patient
  * History of uncontrolled endocrine disorders
  * Physical handicaps that hinder proper oral hygiene
  * Use of experimental devices or drugs within 30 days prior to implant placement surgery
  * Alcoholism or drug abuse
  * Smokers of> 10 cigarettes per day or the equivalent cigar or> 10 tobacco-based chewings per day
  * Conditions or circumstances that prevent the completion of participation in the study or interfere with the analysis of the study results

Local exclusion conditions:

* Local inflammation, including untreated periodontitis
* Patients with erosive lichen planus
* History of local radiation therapy
* Presence of bone lesions
* Unhealed extraction sites
* History of bone reconstruction and bone grafting techniques in the sites where the implants are to be inserted
* Bruxism
* Bleeding index> 30% and number of pockets> 5mm greater than 10

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2021-10-18 (Actual); Primary Completion 2023-06-01 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
Widht of Keratinized mucosa | 2-4-8-12-24 weeks - 1-2-3-4-5 years
  variation of keratized mucosa from t0

SECONDARY OUTCOMES:
implant survival | 1-2-3-4-5 years
  Implant in function
marginal bone loss | 1-2-3-4-5 years
  variation of marginal bone loss over time
Vas Scale | 2 weeks
  Prom: patient VAS scale for post-operative pain, from 0 to 10, where 10 is higher and 0 is minimum.

OTHER OUTCOMES:
Time | day 1
  surgical time differences between the two groups
prosthetic complications | 1-2-3-4-5 years
  number and type of prosthetic complications over time

CONTACTS AND LOCATIONS:
Locations (1):
- Clinica Odontoiatrica Giorgio Vogel, Milan, MI, Italy

IPD SHARING:
Plan to Share IPD: Undecided